CLINICAL TRIAL: NCT05394480
Title: Stress Level Among Dentists In Performing Treatment In Clinic, Deep Sedation, and General Anesthesia
Brief Title: Stress Level Among Dentists in Performing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, esra kizilci, Assist prof dr. Erciyes University pediatric dentistry department, TC Erciyes University
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 82021
Record Dates: First submitted 2022-01-02; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Stress, Job
Keywords: DEEP SEDATION; GENERAL ANESTHESIA; pediatric dentistry; STRESS LEVELS
MeSH Terms: conditions — Occupational Stress | interventions — Blood Pressure; Systole; Diastole

STUDY DESIGN:
Intervention Model Description: In the present study, it was aimed to evaluate the stress which was experienced by dentists working with children while treating children in all three treatment protocols by using objective (salivary cortisol, pulse, blood pressure, O2 saturation) and subjective (Dentists' Stress Questionnaire) findings 27. The H0 hypothesis of the study is that the stress levels of dentists change according to the different treatment protocols.
  each dentist treated 27 patients in 3 different treatment approaches, and the study resulted in a total of 108 patients.
Who Masked: Participant, Care Provider
Masking Description: 4 dentist treated 27 patients in 3 different treatment groups, and the study resulted in a total of 108 patients.
  Children were grouped after being evaluated by a single pediatric dentist. The patients were randomly distributed to the physicians, and their treatment was carried out. The study did not include children with general health problems or whose parents refused to be treated with general anaesthesia/sedation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- clinical treatment (Experimental): 4 dentist treated 36 patient in clinical group
  - For treatment in a clinic, children with positive or definitely positive (Frankl 3 and 4) behaviour according to the Frankl Scale (Behavior Evaluation Scale) 28, with the data observed in the first session, were included in the clinical treatment group. According to the clinical examination of these patients, 36 healthy children aged 5-6 years who did not require pulpal treatment and whose caries level was 1-4 according to the ICDAS (International Caries Detection And Assessment System) 29 scoring were selected. The limits of the treatment were determined as compomer filling applied to 2 primary molars after local anaesthesia, and the duration of the treatment was limited to 30 to 60 minutes.
  Interventions: Diagnostic Test: Blood pressure (Systolic, Diastolic), Pulse value, O2 saturations were measured.
- deep sedation (Experimental): 4 dentist treated 36 patient in clinical group
  - Children aged 48-72 months, children with negative or absolutely negative behaviour (Frankl 1 and 2) according to the Frankl Scale, were reserved for treatment under deep sedation. In order to provide standardization among patients suitable for sedation, 36 children (n=9) whose dmft (decayed, missing, filled teeth index) were less than their age, and the duration of the procedure would be limited to between 30 and 40 minutes, were included in the study.
  Interventions: Diagnostic Test: Blood pressure (Systolic, Diastolic), Pulse value, O2 saturations were measured.
- general anaesthesia (Experimental): 4 dentist treated 36 patient in clinical group
  - Children aged 48-72 months, children with negative or definitely negative behaviour according to the Frankl Scale (Frankl 1 and 2), were reserved for treatment under general anaesthesia. In order to provide standardization among patients suitable for general anaesthesia, 36 healthy children (n=9) whose dmft was equal to, or higher than their age were allocated. In addition, patients whose treatment time would be limited to 30 to 60 minutes were included.
  Interventions: Diagnostic Test: Blood pressure (Systolic, Diastolic), Pulse value, O2 saturations were measured.

INTERVENTIONS:
Diagnostic Test: Blood pressure (Systolic, Diastolic), Pulse value, O2 saturations were measured. — Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit.
  Other Names: Salivary cortisol

SUMMARY:
Purpose: To evaluate the stress levels of dentists working under clinical, deep sedation, or general anaesthesia. Methods: Blood pressure (Systolic, Diastolic blood pressure), Pulse value, O2 saturations were measured, and saliva samples were taken by the dentists 10 minutes before the dental treatment, at the 25th minute of the treatment, and 30 minutes after the treatment under clinic, deep sedation, and general anesthesia. Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit. The data are analayse statistically

DETAILED DESCRIPTION:
Occupational stress, defined as when the resources of the individual are not sufficient to cope with the needs of a situation, is a leading modern health and safety challenge 2.

Although stress is defined as a feeling of tension and pressure, small amounts of stress can be helpful for the individual to cope with difficult situations. The dentist who wants to provide the best treatment for the patient can feel stress and uneasiness when the current conditions are inappropriate. If this stress of dentist is very the desired amount, it can lead to harmful results for patient health.

Especially in pediatric dentistry, behaviour management problems in children, parents' expectations, and behaviours can be more stressful and exhausting in practice. A dentist' s fear and anxiety in children can create various difficulties for the child, parents, dentists, and their team.

Deep sedation is the method in which consciousness is suppressed in a controlled manner by the drug applied, partial loss of protective reflexes, and the response to verbal stimuli is removed. General anaesthesia, on the other hand, is a condition in which the level of patient unconsciousness can be controlled, the patient's protective reflexes are partially or wholly lost, he cannot protect the airway independently, and cannot respond to verbal commands or physical stimuli. Ensuring and maintaining airway patency is vital in sedation applications. In anaesthesia applications, deep sedation in dental procedures is challenging due to the anatomical proximity of the surgical area to the airway, the risk of microaspiration. Dental treatment with general anaesthesia is seen that it is a stressful situation for the practitioner since some complications such as neurological damage, cardiac and respiratory arrest, and even death may occur.

In healthy individuals, stimulation of the sympathetic nervous system at the beginning of the stress response begins with the secretion of epinephrine and norepinephrine from the adrenal medulla. For this reason, sympathetic activity is measured by various evaluation methods such as heart rate, blood pressure, O2 saturation. Salivary cortisol has been accepted as a reliable biomarker of the Hypothalamus-Pituitary-Adrenal system as a delayed stress response.

In the literature review, very few studies investigated occupational stress related to pediatric dentistry. Furthermore, no study was found in which the stress situation in three treatment protocols was evaluated and compared. It was aimed to evaluate the stress which was experienced by dentists working with children while treating children in all three treatment protocols by using objective tests. The H0 hypothesis of the study is that the stress levels of dentists change according to the different treatment protocols.

METHODS This study was approval required for the study was obtained by the clinical research ethics committee from University (No: 82021/32) and conducted following the principles of the Declaration of Helsinki. Both the parents and their children and dentists who agreed to participate in the study provided informed consent.

According to the power analysis, the estimated number of samples was determined as 9 patients in each groups (α error 0.05 and 1-β=0.80). Therefore, each dentist treated 27 patients in 3 different treatment approaches, and the study resulted in a total of 108 patients.Blood pressure (Systolic, Diastolic blood pressure), Pulse value, O2 saturations were measured, and saliva samples were taken by the dentists 10 minutes before the dental treatment, at the 25th minute of the treatment, and 30 minutes after the treatment for all 3 treatment approaches The Saliva Swab Sample Collection kit was used to collect saliva samples. It was placed under the tongue for 2 minutes and was ensured that the swab absorbed the saliva. Afterwards, the swab was centrifuged and placed in saliva storage tubes with a perforated chamber for separating saliva and remaining dry swab. Samples were centrifuged at 3000 rpm for 15 minutes, saliva was cleared of debris and poured to the bottom of the storage tube. Then, saliva in the plastic saliva storage tube was stored at -80 ºC in an upright position until measurements were made 30. After the saliva samples were thawed at room temperature on the day of the measurements, they were taken to the University Medical Faculty Central Biochemistry Laboratory for analysis.

Salivary Cortisol Measurement Protocol:

Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit (Roche Diagnostics GmbH; Mannheim, Germany).

10 µL of sample is incubated with cortisol-specific biotinylated antibody and cortisol derivative labelled with ruthenium complex. Depending on the analyte concentration in the sample and the formation of the respective immune complex, the labelled antibody binding site is filled partly with the sample analyte and partly with the ruthenium hapten.

After streptavidin-coated microparticles have been added, biotin and streptavidin interact. The complex becomes bound to the solid phase.

The reaction mixture is aspirated into the measuring cell on the surface of the electrode. The measuring cell is that the microparticles, magnetically, are captured. Unbound substances are then removed with ProCell/ProCell M. Applying voltage to the electrode induces chemiluminescence emission, which is measured with a photomultiplier.

An instrument-specific calibration curve determines results with 2-point calibration and a master curve acquired via the reagent barcode 30.

Statistical analysis In the study, the analyzes were made with the SPSS 25.0 program. On the analysis of data, descriptive statistics are presented with mean and standard deviation values. In the study, the Kruskal Wallis test was performed to examine the differences in measurements according to dentists and treatment approaches. Mann Whitney U test was used to reveal the evaluation that caused the difference. The Friedman test was used to examine the differences between the measurements in the treatment approaches before, during, and after the procedure.

Results When the findings are evaluated according to the measurement times: systolic and diastolic blood pressure measurements for all dentists before the procedure are similar in clinical, general anaesthesia, and sedation (p>0.05). During the procedure, both systolic and diastolic blood pressure measurements were found to be higher under the deep sedation (p<0.05). It was determined that systolic blood pressure measurements did not differ according to under clinical, general anaesthesia, and deep sedation after the procedure (p>0.05), but diastolic blood pressure measurements differed according to treatment approaches. The measurements under the deep sedation were higher than the clinical and general anaesthesia (p<0.05). Pulse and oxygen saturation measurements before, during, and after the treatment did not differ under clinical, general anaesthesia, and deep sedation. It was observed that cortisol measurements before and during the treatment were not at different levels compared to clinical, general anaesthesia, and deep sedation (p>0.05). After the procedure, cortisol measurements under the deep sedation were higher than clinical and general anaesthesia (p<0.05).

It was observed that the heart rate measurements were at similar levels before, during, and after the procedure under clinical and general anaesthesia. Under the deep sedation, it was determined that the heart rate measurements during the procedure were at higher levels than before and after the procedure (p<0.05).

When authors evaluated the oxygen saturation measurements, the oxygen saturation during the procedure was lower than before and after the procedure.

Cortisol measurements were found to be at different levels according to the processing times in Table 2.

ELIGIBILITY:
Inclusion Criteria:

* 4 dentists, who started their specialization training, simultaneously in Erciyes University Faculty of Dentistry, Department of Pediatric Dentistry, with equal clinical experience and training.
* Woman
* Between the ages of 30-33
* Weights 52-55 kg
* No systemic disease
* Dentists who have actively treated patients for at least 2 years in a clinic, with deep sedation and general anaesthesia are included.

Exclusion Criteria:

* Children who were previously hospitalized due to health problems or who did not live with their biological family were also excluded from the study.

Ages: 30 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | saliva samples were taken by the dentists 10 minutes before the dental treatment
  Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit.
Salivary cortisol | saliva samples were taken by the dentists at the 25th minute of the treatment
  Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit.
Salivary cortisol | saliva samples were taken by the dentists at the 30 minutes after the treatment
  Salivary cortisol was measured by electrochemiluminescence (ECLIA) method using the Cobas Cortisol ll kit.

SECONDARY OUTCOMES:
Systolic, Blood pressure | Systolic Blood pressure were measured by the dentists 10 minutes before the dental treatment
  Systolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)
Diastolic Blood pressure | Diastolic Blood pressure were measured by the dentists 10 minutes before the dental treatment
  Diastolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)
Systolic Blood pressure | Systolic Blood pressure were measured by the dentists at the 25th minute of the treatment
  Systolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)
Diastolic Blood pressure | Diastolic Blood pressure were measured by the dentists at the 25th minute of the treatment
  Diastolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)
Systolic Blood pressure | Systolic Blood pressure were measured by the dentists 30 minutes after the treatment
  Systolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)
Diastolic Blood pressure | Diastolic Blood pressure were measured by the dentists 30 minutes after the treatment
  Diastolic Blood pressure were measured with Automatic Wrist Blood Pressure Monitor, as (mmHg)

OTHER OUTCOMES:
Pulse value | Pulse value were measured by the dentists 10 minutes before the dental treatment
  Pulse value were measured, with Braun YK-81CEU Pulse oximeter, as PRbpm
Pulse value | Pulse value were measured by the dentists at the 25th minute of the treatment
  Pulse value were measured, with Braun YK-81CEU Pulse oximeter, as PRbpm
Pulse value | Pulse value were measured by the dentists 30 minutes after the treatment
  Pulse value were measured, with Braun YK-81CEU Pulse oximeter, as PRbpm
O2 saturations | O2 saturations were measured by the dentists at the 25th minute of the treatment
  O2 saturations were measured with with Braun YK-81CEU Pulse oximeter, SpO2, %
O2 saturations | O2 saturations were measured by the dentists 30 minutes after the treatment
  O2 saturations were measured with Braun YK-81CEU Pulse oximeter, SpO2, %
O2 saturations | Pulse value were measured by the dentists 10 minutes before the dental treatment
  O2 saturations were measured with Braun YK-81CEU Pulse oximeter, SpO2, %

CONTACTS AND LOCATIONS:
Overall Officials: ESRA KIZILCI, 1, Study Chair — erciyes university pediatric dentistry
Locations (1):
- Esra Kizilci, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The raw data are available in the authors

REFERENCES:
- [Background] Basu S, Qayyum H, Mason S. Occupational stress in the ED: a systematic literature review. Emerg Med J. 2017 Jul;34(7):441-447. doi: 10.1136/emermed-2016-205827. Epub 2016 Oct 11. PMID 27729392